CLINICAL TRIAL: NCT03389464
Title: Computer-based Treatment of Dysfunctional Beliefs in Depressive Inpatients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Regensburg (Other)
Collaborators: Klinik und Poliklinik für Psychiatrie und Psychotherapie der Universität Regensburg am Bezirksklinikum Regensburg, Germany (Unknown)
Responsible Party: Principal Investigator, Shiban Youssef, Principal Investigator, University of Regensburg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Face
Record Dates: First submitted 2017-12-14; First posted 2018-01-03 (Actual); Last update posted 2018-05-02 (Actual); Status verified 2018-05

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- confrontation group (Experimental): computer-based confrontation with dysfunctional beliefs
  Interventions: Behavioral: computer-based confrontation with dysfunctional beliefs
- control group (No Intervention): no computer-based confrontation with dysfunctional beliefs

INTERVENTIONS:
Behavioral: computer-based confrontation with dysfunctional beliefs — Patients will be presented with a virtual agent confronting them with their dysfunctional core beliefs (e.g. "You are worthless"). Participants will be instructed to contradict these virtual agents (e.g. "That's not true, I'm a wonderful person").
  Arms: confrontation group

SUMMARY:
The aim of the present study is to investigate whether confronting depressive patients with their dysfunctional core beliefs via a computer program results in a reduction of the patients' dysfunctional beliefs. Patients will be presented with a virtual agent confronting them with their dysfunctional core beliefs (e.g. "You are worthless"). Participants will be instructed to contradict these virtual agents (e.g. "That's not true, I'm a wonderful person").

DETAILED DESCRIPTION:
The aim of the present study is to investigate whether confronting depressive patients with their dysfunctional core beliefs via a computer program results in a reduction of the patients' dysfunctional beliefs. Participants will randomly be assigned to the experimental or control group. In the course of the study, experimental participants will be presented with a virtual agent confronting them with their dysfunctional core beliefs (e.g. "You are worthless"). Experimental participants will be instructed to contradict these virtual agents (e.g. "That's not true, I'm a wonderful person").

A group of inpatients (male/female) suffering from depression will participate in the study. The patients will be recruited at the "Klinik und Poliklinik für Psychiatrie und Psychotherapie der Universität Regensburg am Bezirksklinikum Regensburg".

The study will be divided into five sessions taking place on consecutive days. Furthermore, there will be a follow-up.

Session 1:

In the course of this session participants will be informed about the experimental procedure and sign an informed consent. Exclusion criteria will be assessed via self-report and by consulting the responsible therapist. Participants will be asked to fill in the German version of the Beck Depression Inventory-II and German version of the Dysfunctional Attitude Scale. The experimenter will explain the concept of dysfunctional "core beliefs" to the participants and give examples. Participants will be asked to write down three individual core beliefs (e.g. "I'm worthless") and to rate how much they believe in each of these three core beliefs (on a scale ranging from 0% to 100%). Furthermore, participants will be asked to write down alternative beliefs for each of the three core beliefs and to rate (on a scale ranging from 0% to 100%) how much they believe in these alternative beliefs.

Sessions 2 to 4 (intervention):

During these sessions, the experimental participants will be seated in front of a computer. The experimenter will read aloud the participants' core beliefs with the virtual agent on the computer screen moving his lips accordingly. Thus, participants will get the impression of the agent speaking to them. Participants will be instructed to contradict the agent. There will be 10 trials per core belief (30 trials per session, 90 trials in total). At the end of each session, participants will be asked to rate how much they believe in each of their core beliefs as well as in each of their alternative beliefs. Furthermore, they will be asked to rate (on a scale ranging from 0% to 100%) how hard it was for them to contradict the virtual agent. Control subjects will not undergo sessions 2 to 4.

Session 5:

Participants will fill in the German version of the Beck Depression Inventory-II and the German version of Dysfunctional Attitude Scale and give a conviction rating for each of their three core beliefs and each of their alternative beliefs.

Follow-up (after two weeks):

Participants will fill in the German version of the Beck Depression Inventory-II and the German version of the Dysfunctional Attitude Scale and give a conviction rating for each of their three core beliefs and each of their alternative beliefs.

ELIGIBILITY:
Inclusion Criteria:

• diagnosis of a depressive disorder

Exclusion Criteria:

* substantial and imminent suicide risk
* current psychotic symptoms
* history of psychotic symptoms
* current manic episode
* current diagnosis of alcohol or drug abuse or dependence
* hearing problems
* poor eyesight
* pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-01-08 (Actual); Primary Completion 2018-09-27 (Estimated); Study Completion 2018-09-27 (Estimated)

PRIMARY OUTCOMES:
change in the score on the Dysfunctional Attitude Scale | at baseline, one day after the end of the intervention, at follow-up (2 weeks after the end of the intervention)
  change in the score (ranging from 40 to 280 with higher scores indicating more dysfunctional attitudes) on the German version of the Dysfunctional Attitude Scale

SECONDARY OUTCOMES:
change in the conviction ratings for the dysfunctional beliefs | at baseline, one day after the end of the intervention, at follow-up (2 weeks after the end of the intervention)
  Participants will be asked to rate (on a scale ranging from 0% to 100%) how much they belief in their dysfunctional beliefs
change in the conviction ratings for the alternative beliefs | at baseline, one day after the end of the intervention, at follow-up (2 weeks after the end of the intervention)
  Participants will be asked to rate (on a scale ranging from 0% to 100%) how much they belief in their alternative beliefs
change in the score on the Beck Depression Inventory-II | at baseline, one day after the end of the intervention, at follow-up (2 weeks after the end of the intervention)
  change in the score (ranging from 0 to 63 with higher scores indicating more severe depressive symptoms) on the German version of the Beck Depression Inventory-II

OTHER OUTCOMES:
change in the conviction ratings for the dysfunctional beliefs (exerimental participants only) | at baseline, on the first day of the intervention, on the second day of the intervention, on the third day of the intervention, one day after the end of the intervention, at follow-up (2 weeks after the end of the intervention)
  Experimental participants will be asked to rate (on a scale ranging from 0% to 100%) how much they belief in their dysfunctional beliefs
change in the conviction ratings for the alternative beliefs (exerimental participants only) | at baseline, on the first day of the intervention, on the second day of the intervention, on the third day of the intervention, one day after the end of the intervention, at follow-up (2 weeks after the end of the intervention)
  Experimental participants will be asked to rate (on a scale ranging from 0% to 100%) how much they belief in their alternative beliefs
change in the difficulty ratings (experimental participants only) | on the first day of the intervention, on the second day of the intervention, on the third day of the intervention
  Experimental participants will be asked to rate (on a scale ranging from 0% to 100%) how hard it was for them to contradict the virtual agent

CONTACTS AND LOCATIONS:
Overall Officials: Youssef Shiban, Prof., Principal Investigator — PFH - Private University of Applied Sciences
Locations (1):
- medbo Bezirksklinikum Regensburg, Regensburg, Germany

REFERENCES:
- [Background] Beck AT, Steer RA, Brown GK. Beck Depression Inventory - Second Edition. Manual. San Antonio, TX: The Psychological Corporation, 1996.
- [Background] Hautzinger M, Keller F, Kühner C. BDI-II - Beck Depressions-Inventar - Manual. Frankfurt: Harcourt Test Services, 2006.
- [Background] Hautzinger M, Joormann J, Keller F. DAS - Skala dysfunktionaler Einstellungen - Manual. Göttingen: Hogrefe, 2005.
- [Background] Weissman AN, Beck AT. Development and validation of the Dysfunctional Attitude Scale: A preliminary investigation. Paper presented at the annual meeting of the Association for the Advancement of Behavior Therapy, Chicago, 1978.